CLINICAL TRIAL: NCT04178616
Title: Assessment of the Prevalence of Olfactory Disorders in Systemic Scleroderma
Acronym: SCLEROLF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Following the COVID-related health crisis, nasofibroscopic sampling could no longer be carried out
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018_84; 2019-A01083-54 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2019-09-30; First posted 2019-11-26 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Olfactory Disorders; Scleroderma
MeSH Terms: conditions — Scleroderma, Diffuse

STUDY DESIGN:
Intervention Model Description: The study is single-group epidemiologic study, without any control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- systemic sclerosis patients population (Other): All the patients with systemic sclerosis disease followed in day-care in a tertiary hospital are eligible to be enrolled in the study.
  Interventions: Diagnostic Test: olfactory testing with specific odorants (localisation and identification)

INTERVENTIONS:
Diagnostic Test: olfactory testing with specific odorants (localisation and identification) — Olfactory testing : ETOC (European Test of Olfactory capabilities)
  Other Names: nasofibroscopy to identify sinonasal mucosa diseases

SUMMARY:
Prospective monocentric study of patients with systemic sclerosis disease.

The primary outcome is to define the prevalence of olfactory disorders (hyposmia and anosmia) in systemic sclerosis disease.

The secondary outcomes are:

* To assess the correlation of olfaction disorders with clinical and biological and factors related to systemic sclerosis patients.
* To estimate the frequency of sinonasal disorders in patients with systemic sclerosis disease

ELIGIBILITY:
Inclusion Criteria:

* Men and/or women
* With systemic sclerosis disease
* Patient willing to comply with all procedures of the study and its duration
* Social insured patients

Exclusion Criteria :

* Patient with medical history of chronic rhinosinusitis (CRS), previously known for olfactory disorders secondary to another etiology (skull base trauma, viral rhinosinusitis)
* Past history of sinonasal surgery
* Patient unable to receive informed information
* Refusal to sign the consent form
* Unwillingness or inability to follow the study procedures, in the opinion of the investigator
* Person deprived of the liberty
* Non-coverage by the social security insurance
* Person benefiting from a system of legal protection (guardianship…)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2019-12-31 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
Percentage of patient with hyposmia defined by a ETOC (European Test of Olfactory Capabilities) score strictly inferior to 27 points | once time, Baseline
  The European Test of Olfactory Capabilities is an olfactory test based on standardized odorants.A composite score evaluates the ability of the patients to define odors localisation and odors identification.The maximum global score is 32 points, the minimum is 0 point. The localisation ability score is rated from 0 to 16 points; The identification score is rated from 0 to 16 points. An hyposmia is defined by a global score strictly inferior to 27 points.

SECONDARY OUTCOMES:
Percentage of patient with anosmia defined by a ETOC (European Test of Olfactory Capabilities) score strictly inferior to10 points | once time, Baseline
  The European Test of Olfactory Capabilities is an olfactory test based on standardized odorants. A composite score evaluates the ability of the patients to define odors localisation and odors identification. The maximum global score is 32 points, the minimum is 0 point. The localisation ability score is rated from 0 to 16 points; The identification score is rated from 0 to 16 points. An anosmia is defined by an global score strictly inferior to 10 points.
Percentage of patients with an unilateral Lund Kennedy score of more than 3 points. | once time, Baseline
  Evaluation of nasal mucosa inflammation status is based on Lund-Kennedy endoscopic score. The Lund Kennedy score ranged from 0 to 8 points for each nasal fossa. It evaluates oedema, discharge, the presence of polyps and crusting, that can be seen through nasal fibroscopy. A score strictly under 3 points on each side is considered as non pathologic whereas a score equal or over 3 points on each side is pathological. A higher score means a worse outcome.
Measurement of systemic sclerosis disease activity with Medsger Score | once time, Baseline
  Medsger Score estimates disease involvement of each organ (heart, vessels, skin, brain, kidney, gut, muscle, joint and loss of weight,) ranging from 0 to 4 (0: normal, 1: mild, 2: moderate, 3: severe, 4: terminal). The score ranges from 0 to 36 points.A higher score means a worse outcome.
Correlation between global olfactory score measured with ETOC score and systemic sclerosis disease activity measured with Medsger Score | once time, Baseline
  The ETOC score ranges from 0 to 32 points ( as previously described ).A higher score means a better outcome.
  Medsger score ranges from 0 to 36 points. A higher score means a worse outcome.
Correlation between global olfactory score measured with ETOC score and skin involvement severity measured with Rodnan score. | once time, Baseline
  The ETOC score ranges from 0 to 32 points ( as previously described ). A higher score means a better outcome.
  The Rodnan score measured skin thickness (0 : normal, 1 : mild, 2: moderate, 3: severe) on 17 different sites. A global score between 0 point to 51 points is established.A higher score means a worse outcome
Correlation between global olfactory score measured with ETOC score and systemic sclerosis disease activity measured with Health Assessment Questionnaire (HAQ) score | once time, Baseline
  The ETOC score ranges from 0 to 32 points (as previously described ). A higher score means a better outcome.
  The Health Assessment Questionnaire is based on 20 questions related to routine activities with a grading system ranging from 0 to 3 (0: no difficulty, 1: moderate difficulty, 2: severe difficulty, 3: total incapacity). A global score between 0 point to 60 points is established. a higher HAQ score means a worse outcome
Correlation between global olfactory score measured with ETOC score and the rhinologic quality of life score measured with the sinonasal outcome test 22) | once time, Baseline
  The ETOC score ranges from 0 to 32 points ( as previously described ). A higher score means a better outcome.
  The sinonasal outcome test 22 is based on 22 questions with a grading from 0 to 5 ( 0: no probem, 1: very mild problem, 2: mild problem, 3: moderate problem, 4: severe problem, 5: very severe problem). A global score between 0 and 110 points is measured. A higher score means a worse outcome.
Correlation between global olfactory score measured with ETOC and Hospital anxiety and Depression (HAD) scale. | once time, Baseline
  The ETOC score ranges from 0 to 32 points ( as previously described ). A higher score means a better outcome.
  The Hospital anxiety and Depression (HAD) scale is based on 14 questions with a grading system ranging from 0 to 3. A global score between 0 and 42 is measured. A higher score means a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: David Launay, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Claude Huriez Chu Lille, Lille, France

REFERENCES:
- [Background] Amital H, Agmon-Levin N, Shoenfeld N, Arnson Y, Amital D, Langevitz P, Balbir Gurman A, Shoenfeld Y. Olfactory impairment in patients with the fibromyalgia syndrome and systemic sclerosis. Immunol Res. 2014 Dec;60(2-3):201-7. doi: 10.1007/s12026-014-8573-5. PMID 25424576
- [Result] Bombini MF, Peres FA, Lapa AT, Sinicato NA, Quental BR, Pincelli ASM, Amaral TN, Gomes CC, Del Rio AP, Marques-Neto JF, Costallat LTL, Fernandes PT, Cendes F, Rittner L, Appenzeller S. Olfactory function in systemic lupus erythematosus and systemic sclerosis. A longitudinal study and review of the literature. Autoimmun Rev. 2018 Apr;17(4):405-412. doi: 10.1016/j.autrev.2018.02.002. Epub 2018 Feb 11. PMID 29444467